CLINICAL TRIAL: NCT01339468
Title: A Phase IV, Randomized, Open-label, Comparative, Single-center Study to Assess the Pharmacokinetics, Safety and Efficacy of Advagraf® (Modified Release Tacrolimus) and Prograf® (Tacrolimus) in de Novo Living Donor Liver Transplant Recipients
Brief Title: A Study to Assess the Pharmacokinetics, Safety and Efficacy of Advagraf and Prograf in de Novo Liver Transplantation
Acronym: MAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR-08-04-KOR_Main
Record Dates: First submitted 2011-04-12; First posted 2011-04-20 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Liver Transplantation
Keywords: advagraf; prograf; living donor liver transplantation; FK506; Immunosuppressant
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Intravenous Prograf therapy followed by oral Advagraf therapy
  Interventions: Drug: Advagraf; Drug: Prograf
- Arm 2 (Active Comparator): Intravenous Prograf therapy followed by oral Prograf therapy
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: Advagraf — oral
  Other Names: FK506E; modified release tacrolimus
  Arms: Arm 1
Drug: Prograf — oral
  Other Names: FK506; tacrolimus
  Arms: Arm 2
Drug: Prograf — intravenous
  Other Names: tacrolimus; FK506

SUMMARY:
The purpose of this study is to investigate and compare the pharmacokinetic parameters of tacrolimus from Advagraf and Prograf in de nove living donor liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* subject receiving a primary, partial liver graft from a living donor
* subject must receive the first dose of tacrolimus and corticosteroids after operation and are expected to be maintained on tacrolimus throughout the study. MMF could be combined

Exclusion Criteria:

* subjects receiving a multi-organ transplant or having previously received an organ transplant (including liver re-transplantation)
* subjects receiving an auxiliary graft or in whom a bio-artificial liver (cell system) has been used
* subjects allergic or intolerant to macrolide antibiotics or tacrolimus
* subjects requiring immunosuppressive treatment and / or systemic chemotherapy prior to transplantation
* subjects with malignancies or a history of malignancy within the last 5 years, with the exception of those with basalioma or squamous cell carcinoma of the skin
* subjects with systemic infection requiring treatment, except viral hepatitis
* subjects with severe diarrhoea, vomiting, active peptic ulcer or gastrointestinal disorder that may affect the absorption of tacrolimus
* subjects with serum creatinine > 1.5mg/dl
* subjects taking or having taken potassium preserved diuretics
* subjects with any form of substance abuse, psychiatric disorder or condition which, in the opinion of the investigator, may complicate communication with the investigator
* subjects participating or having participated in another clinical trial and/or those taking or having taken an investigational / non-registered drug in the past 28 days
* subjects or donors known to be HIV positive
* donors known to be HBV, HCV positive and/or IgM positive of CMV, EBV

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04-27 (Actual); Primary Completion 2014-05-27 (Actual); Study Completion 2014-05-27 (Actual)

PRIMARY OUTCOMES:
AUC0-24 (Area under the curve for 24 hours) of tacrolimus plasma concentration | Day 6 and day 21

SECONDARY OUTCOMES:
Cmax (maximum concentration) of tacrolimus plasma concentration | Day 6 and day 21
Incidence of the composite event: graft loss (defined as re-transplantation or death) or biopsy confirmed acute rejection (BCAR) | up to 24 weeks
Time to first incidence of the composite event: graft loss (defined as re-transplantation or death) or biopsy confirmed acute rejection (BCAR) | up to 24 weeks
Safety assessed by the incidence of adverse events and lab-tests | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Seoul, South Korea

REFERENCES:
- [Derived] Shin MH, Song GW, Lee SG, Hwang S, Kim KH, Ahn CS, Moon DB, Ha TY, Jung DH, Park GC, Yun YI, Kim WJ, Kang WH, Kim SH, Jiang H, Lee S, Tak EY. Once-daily, prolonged-release tacrolimus vs twice-daily, immediate-release tacrolimus in de novo living-donor liver transplantation: A Phase 4, randomized, open-label, comparative, single-center study. Clin Transplant. 2018 Sep;32(9):e13376. doi: 10.1111/ctr.13376. Epub 2018 Aug 26. PMID 30098071
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=131
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=130